CLINICAL TRIAL: NCT04800393
Title: The Impact of Inhalation vs Total Intravenous Anesthesia on the Immune Status and Mortality in Patients Undergoing Breast Cancer Surgery: a Prospective Double-Blind Randomized Clinical Trial (TeMP - Trial).
Brief Title: The Impact of Inhalation vs Total Intravenous Anesthesia on the Immune Status and Mortality in Patients Undergoing Breast Cancer Surgery: a Prospective Double-Blind Randomized Clinical Trial.
Acronym: TeMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow Clinical Scientific Center (Other)
Collaborators: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Principal Investigator, Valerii Subbotin, PhD, Moscow Clinical Scientific Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TeMP 2021
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; Breast Cancer
Keywords: Anesthesia; Breast Cancer; Phagocyte Cell Dysfunction; Immune Suppression; Inhalation anesthesia; volatile anesthesia; total intravenous anesthesia; interleukins; phagocytosis; neutrophil-lymphocyte ratio; natural killers; oncology
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalation anesthesia (Experimental)
  Interventions: Drug: Sevoflurane
- Total intravenous anesthesia (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — induction of anesthesia with propofol, maintenance of anesthesia with sevoflurane during breast cancer surgery
  Arms: Inhalation anesthesia
Drug: Propofol — propofol-based total intravenous anesthesia during breast cancer surgery
  Arms: Total intravenous anesthesia

SUMMARY:
Even decade ago it was believed that the choice method of anesthesia did not affect the course of the oncological process, but recent evidence has begun to emerge that inhalation anesthesia vs TIVA is associated with a higher number of adverse outcomes. Apparently, it makes sense to conduct mRCT in order to assess the effect of IA on immune system in patients operated on for breast cancer comprehensively. The results of that kind of RCT may finally give us an answer whether the choice of anesthesia affects the immune status of patients undergoing surgery for breast cancer. The evaluation of complications and long-term survival will allow to recommend to use or not to use IA for this type of surgery.

Objective: The Impact of Inhalation vs Total Intravenous Anesthesia on the Immune Status and Mortality in Patients Undergoing Breast Cancer Surgery

DETAILED DESCRIPTION:
The power calculation for this study was based on an assessment of Neutrophil-lymphocyte ratio (NLR) in patients undergoing breast cancer resection with total intravenous and inhalation anesthesia in two studies:

1. Cho J.S. et al., 2017 - 48 patients (PMID: 28924368, TIVA group: NLR = 3.37 ± 1.27; inhalation group: NLR = 3.85 ± 1.46)
2. Ní Eochagáin A. et al., 2018 - 116 patients (PMID: 29457215, TIVA group: NLR = 3.20 ± 1.37; inhalation group: NLR = 4.10 ± 1.90).

The pooled mean NLR in the TIVA group is 3.25±1.34, in the inhalation anesthesia group: 4.03±1.78.

Difference in means (effect size): 0.78, for level α=0.05, power 1-β=80% and expected standard deviation of 1.5, 65 patients in each group should be recruited, taking into account a 10% margin (total number of patients: 130).

ELIGIBILITY:
Inclusion Criteria:

* The age of the patients is from 45 to 74 years;
* Primary operable breast cancer (BC) without prior chemotherapy;
* Cytologically confirmed breast malignant tumor of IA-IIA stages (T1-2, N0, M0);
* Signed informed consent.

Exclusion Criteria:

* Acute cerebrovascular accident (CVA) occurred in the previous 6 months;
* Myocardial infarction (MI) occurred in the previous 6 months;
* Acute arterial thrombosis occurred in the previous 6 months;
* Acute venous thromboembolism occurred in the previous 6 months;
* Subarachnoid hemorrhage occurred during the previous 3 months;
* Chronic kidney disease (CKD) stage 3B-5;
* Сhronic heart failure (NYHA) class 3-4;
* Pregnancy;
* History of another location cancer;
* History of drug addiction;
* Autoimmune diseases in history;
* Post-randomization: withdrawal of informed consent (refusal to continue participating in the study);
* Post-randomization: surgical intervention, performed not in full (verified non-resected lesions in the early p/o period, 2 weeks p/o).

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Neutrophil-lymphocyte ratio | 1 hour after surgery
  Absolute number of neutrophils divided by the absolute number of lymphocytes
Neutrophil-lymphocyte ratio | 24 hours after surgery
  Absolute number of neutrophils divided by the absolute number of lymphocytes

SECONDARY OUTCOMES:
Matrix metallopeptidase 9 | 1 hour after surgery
  ng/mL
Matrix metallopeptidase 9 | 24 hour after surgery
  ng/mL
C-reactive protein | 1 hour after surgery
  mg/L
C-reactive protein | 24 hour after surgery
  mg/L
Natural killer cells of blood (CD3-CD16 +) | 1 hour after surgery
  Absolute number (х 10^9 /L)
Natural killer cells of blood (CD3-CD16 +) | 24 hour after surgery
  Absolute number (х 10^9 /L)
Immunoregulatory index of T helpers (CD3 + CD4 +) / cytotoxic T cells (CD3 + CD8 +) | 1 hour after surgery
  the ratio of T helper cells to cytotoxic T cells
Immunoregulatory index of T helpers (CD3 + CD4 +) / cytotoxic T cells (CD3 + CD8 +) | 24 hour after surgery
  the ratio of T helper cells to cytotoxic T cells
IL-6 | 1 hour after surgery
  pg/ml
IL-6 | 24 hour after surgery
  pg/ml

OTHER OUTCOMES:
T cells of blood (CD3 +) | 1 hour after surgery
  Absolute number (х 10 /L)
T cells of blood (CD3 +) | 24 hours after surgery
  Absolute number (х 10^9 /L)
T helpers of blood (CD3 + CD4 +) | 1 hour after surgery
  Absolute number (х 10^9 /L)
T helpers of blood (CD3 + CD4 +) | 24 hours after surgery
  Absolute number (х 10^9 /L)
Cytotoxic T cells of blood (CD3 + CD8 +) | 1 hour after surgery
  Absolute number (х 10^9 /L)
Cytotoxic T cells of blood (CD3 + CD8 +) | 24 hours after surgery
  Absolute number (х 10^9 /L)
B cells of blood (CD19 + CD3-) | 1 hour after surgery
  Absolute number (х 10^9 /L)
B cells of blood (CD19 + CD3-) | 24 hour after surgery
  Absolute number (х 10^9 /L)
T cells (CD3 +) + B cells (CD19 + CD3 -) + Natural killer cells (CD3-CD16 +) of blood | 1 hour after surgery
  percentage
T cells (CD3 +) + B cells (CD19 + CD3 -) + Natural killer cells (CD3-CD16 +) of blood | 24 hours after surgery
  percentage
Phagocytosis | 1 hour after surgery
  percentage
Phagocytosis | 24 hours after surgery
  percentage
IgA | 1 hour after surgery
  g/L
IgA | 24 hours after surgery
  g/L
IgM | 1 hour after surgery
  g/L
IgM | 24 hours after surgery
  g/L
IgG | 1 hour after surgery
  g/L
IgG | 24 hours after surgery
  g/L
Complement component C3 | 1 hour after surgery
  g/L
Complement component C3 | 24 hours after surgery
  g/L
Complement component C4 | 1 hour after surgery
  g/L
Complement component C4 | 24 hours after surgery
  g/L
Overall survival | 1 year
  percentage of survival patients
Overall survival | 3 year
  percentage of survival patients
Overall survival | 5 year
  percentage of survival patients
Disease-free survival | 1 year
  percentage of survival patients
Disease-free survival | 3 year
  percentage of survival patients
Disease-free survival | 5 year
  percentage of survival patients

CONTACTS AND LOCATIONS:
Overall Officials: Valerii Subbotin, PhD, Principal Investigator — Moscow Scientific Clinical Center; Valery Likhvantsev, PhD, Study Director — Negovsky Reanimatology Research Institute
Locations (1):
- Moscow Scientific Clinical Center, Moscow, Russia